CLINICAL TRIAL: NCT00365859
Title: A 52-Week, Open-Label, Multicenter Study of the Safety and Tolerability of Aripiprazole Flexibly Dosed in the Treatment of Children and Adolescents With Autistic Disorder
Brief Title: Study of Aripiprazole in the Treatment of Serious Behavioral Problems in Children and Adolescents With Autistic Disorder (AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-180
Record Dates: First submitted 2006-08-15; First posted 2006-08-18 (Estimated); Results first posted 2010-01-25 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2010-06

CONDITIONS: Autistic Disorder; Behavioral Symptoms
Keywords: Serious behavioral problems in children and adolescents with AD; behavioral problems
MeSH Terms: conditions — Autistic Disorder; Behavioral Symptoms; Problem Behavior | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- De Novo (Experimental): De novo participants (those who did not participate in protocol (CN138-178 [NCT00332241] or CN138-179 [NCT00337571]) assigned to open-label aripiprazole (oral tablet), flexibly dosed (2 to 15 mg/day) taken once daily, started at 2 mg/day on Day 1. Target daily dose was 5 mg, 10 mg, or 15 mg; maximum dose, regardless of weight, was 15 mg. Dose increases were incremental (dose levels are 2 mg, 5 mg, 10 mg, and 15 mg), occurring no more often than every 4 days, and were based on assessment of efficacy and tolerability at the current dose. The dosage could be adjusted downward if the patient experienced intolerance at any time to the current dose.
  Interventions: Drug: Aripiprazole
- Rollover Placebo (Experimental): Participants who completed participation in protocol (CN138-178 [NCT00332241] or CN138-179 [NCT00337571]) on placebo treatment and continued to meet all of the inclusion criteria and none of the exclusion criteria. Assigned in this study to open-label aripiprazole (oral tablet), flexibly dosed (2 to 15 mg/day) taken once daily, started at 2 mg/day on Day 1. Target daily dose was 5 mg, 10 mg, or 15 mg; maximum dose, regardless of weight, was 15 mg. Dose increases were incremental (dose levels are 2 mg, 5 mg, 10 mg, and 15 mg), occurring no more often than every 4 days, and were based on assessment of efficacy and tolerability at the current dose. The dosage could be adjusted downward if the patient experienced intolerance at any time to the current dose.
  Interventions: Drug: Aripiprazole
- Rollover Aripiprazole (Experimental): Participants who completed participation in protocol CN138-178 [NCT00332241] or CN138-179 [NCT00337571] on aripiprazole treatment and continued to meet all of the inclusion criteria and none of the exclusion criteria. Assigned in this study to open-label aripiprazole (oral tablet), flexibly dosed (2 to 15 mg/day) taken once daily, started at 2 mg/day on Day 1. Target daily dose was 5 mg, 10 mg, or 15 mg; maximum dose, regardless of weight, was 15 mg. Dose increases were incremental (dose levels are 2 mg, 5 mg, 10 mg, and 15 mg), occurring no more often than every 4 days, and were based on assessment of efficacy and tolerability at the current dose. The dosage could be adjusted downward if the patient experienced intolerance at any time to the current dose.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 2, 5, 10, or 15 mg, once daily, 52 weeks
  Other Names: Abilify; BMS-337039

SUMMARY:
This study will provide long-term safety data for patients who are taking aripiprazole for up to 1 year. Most patients enrolled in this study will have participated in a short-term study with aripiprazole (CN138-178 [NCT00332241] or CN138-179 [NCT00337571]).

ELIGIBILITY:
Inclusion Criteria - Rollover:

* Completed 8 weeks of treatment in one of the following double-blind clinical trials: CN138-178 [NCT00332241] or CN138-179 [NCT00337571]
* No significant protocol violations and sufficient medical justification to continue on open-label treatment with aripiprazole

Inclusion Criteria - De Novo:

* Meets current Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV TR) diagnostic criteria for AD and demonstrates serious behavioral problems - diagnosis confirmed by Autism Diagnostic Interview-Revised (ADI-R) or the patient meets the current Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV TR) diagnostic criteria for AD and has a history of behavioral problems that are currently being treated with psychotropic medication
* Mental age of at least 18 months
* Male or female 6 to 17 years of age, inclusive, at the time of enrollment

Exclusion Criteria:

* Patients considered treatment resistant to neuroleptic medication based on lack of therapeutic response to 2 different neuroleptics after treatment of at least 3 weeks each
* Patients previously treated and not responding to aripiprazole treatment
* The patient is currently diagnosed with another disorder on the autism spectrum, including pervasive developmental disorder-not otherwise specified (PDD-NOS), Asperger's Disorder, Rett's Disorder, Fragile-X Syndrome or Childhood Disintegrative Disorder
* Current diagnosis of bipolar disorder, psychosis, schizophrenia, or major depression
* A seizure in the past year
* History of severe head trauma or stroke
* Non-pharmacologic therapy (e.g. psychotherapy, behavior modification) should be stable prior to screening and consistent throughout the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- United States (55):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harmonex Neuroscience, Dothan, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Univ of Arizona, Tuscon, Arizona
  - Clinical Innovations, Inc, Costa Mesa, California
  - Peninsula Research Assoc, Rolling Hills Estate, California
  - University Of California-Davis Health Science Center, Sacramento, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Stanford University School Of Medicine, Stanford, California
  - The Children's Hospital, Aurora, Colorado
  - Offices of Gregory Marsella, MD, PA, Boca Raton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Miami Children's Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Children's Developmental Center, Winter Park, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Institute For Behavioral Medicine, Smyrna, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Ladders Clinic, Wellsley, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Children's Hospital Of Michigan, Detroit, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Munroe-Meyer Institute Diagnostic Center, Omaha, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - North Shore - Long Island Jewish Health System, Bethpage, New York
  - Seaver and New York Autism Center of Excellence, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY at Stony Brook - School of Medicine, Stony Brook, New York
  - Mission Hospitals - Mission Children's Clinics, Asheville, North Carolina
  - University of NC, Chapel Hill, North Carolina
  - Duke Child and Family Study Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Nisonger Center, Columbus, Ohio
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - UT Medical Group, Department Of Psychiatry, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - North San Antonio Healthcare Associates, San Antonio, Texas
  - Children's National Medical Center, Fairfax, Virginia
  - Neuroscience, Inc, Herndon, Virginia
  - Monarch Research Associates, Norfolk, Virginia
  - Virginia Treatment Center For Children, Richmond, Virginia
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Autism Spectrum Treatment and Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Marcus RN, Owen R, Manos G, Mankoski R, Kamen L, McQuade RD, Carson WH, Findling RL. Safety and tolerability of aripiprazole for irritability in pediatric patients with autistic disorder: a 52-week, open-label, multicenter study. J Clin Psychiatry. 2011 Sep;72(9):1270-6. doi: 10.4088/JCP.09m05933. Epub 2011 Jul 26. PMID 21813076
- [Derived] Marcus RN, Owen R, Manos G, Mankoski R, Kamen L, McQuade RD, Carson WH, Corey-Lisle PK, Aman MG. Aripiprazole in the treatment of irritability in pediatric patients (aged 6-17 years) with autistic disorder: results from a 52-week, open-label study. J Child Adolesc Psychopharmacol. 2011 Jun;21(3):229-36. doi: 10.1089/cap.2009.0121. PMID 21663425
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: Centers for Disease Control and Prevention (CDC) algorithm for BMI and body weight z-scores — http://www.cdc.gov/growthcharts/percentile_data_files.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 109 participants were enrolled in the De Novo arm, 70 in the Rollover Placebo arm, and 174 in the Rollover Aripiprazole arm. 23 participants in the De Novo arm were considered "baseline failures," and did not enter the treatment phase.
Period: Overall Study
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Started | 86 | 70 | 174 | 330
Safety Population | 86 | 70 | 174 | 330
Efficacy Population | 84 (1 patient was lost to follow-up and 1 not included due to moderate sedation (total=2)) | 69 (1 not included due to increased alanine aminotransferase (ALT) prior to treatment with aripiprazole) | 169 (3 lost to follow-up, 1 not included due to mild increased appetite, 1 to family emergency (total=5)) | 322
Completed | 55 | 37 | 107 | 199
Not Completed | 31 | 33 | 67 | 131

BASELINE CHARACTERISTICS:
Groups:
- De Novo; Rollover Placebo; Rollover Aripiprazole: As previously described in Participant Flow
- Total: Total of all reporting groups
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Age, Customized [Number; unit: participants]
  6 to 12 years | 69 | 56 | 138 | 263
  13 to 17 years | 17 | 14 | 36 | 67
Age Continuous [Mean (Standard Deviation); unit: years] | 9.7 (3.13) | 9.6 (2.95) | 9.5 (3.00) | 9.6 (3.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 19 | 43
  Male | 70 | 62 | 155 | 287

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Emergent Adverse Events (AEs), Deaths, AEs Leading to Discontinuation, Extra Pyramidal Syndrome (EPS)-Related AEs
Description: Participants with Adverse Events (AEs), Deaths, Serious AEs (SAEs), and AEs leading to study discontinuation. AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: From Screening (up to 42 days prior to treatment start) through Week 52 (end of study) for SAEs; from Week 0 (Baseline) through Week 52 (End of Study) for AEs
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Deaths | 0 | 0 | 0 | 0
  Treatment-Emergent SAEs | 3 | 1 | 5 | 9
  Treatment-Emergent AEs | 75 | 63 | 148 | 286
  Treatment-Emergent AEs Leading to Discontinuation | 9 | 10 | 14 | 33
  Treatment-Emergent EPS-Related AEs | 16 | 6 | 26 | 48

2. Primary Outcome: Mean Change From Baseline in Total Simpson-Angus Scale (SAS) At Week 8, Week 26, and Week 52
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50. Negative change scores indicate improvement.
Time Frame: Baseline, Week 8, Week 26, Week 52
Population: Safety Sample - Observed Cases (OC) Data Set and Endpoint - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
units on a scale
  Baseline (n=79, 63, 153, 295) | 10.7 (1.40) | 10.6 (1.17) | 11.0 (2.11) | 10.8 (1.77)
  Change at Week 8 (n=77, 60, 145, 282) | -0.3 (1.13) | 0.1 (1.51) | -0.4 (2.12) | -0.2 (1.78)
  Change at Week 26 (n=61, 47, 126, 234) | -0.2 (1.59) | 0.2 (1.42) | -0.6 (1.96) | -0.3 (1.79)
  Change at Week 52 (n=48, 36, 91, 175) | -0.6 (1.44) | 0.3 (1.80) | -0.5 (1.82) | -0.3 (1.75)
  Change at Endpoint (LOCF) (n=79, 63, 153, 295) | -0.2 (1.70) | 0.3 (1.59) | -0.3 (2.06) | -0.1 (1.89)

3. Primary Outcome: Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) At Week 8, Week 26, and Week 52
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). The AIMS Total Score has a possible range from 0 to 28. Negative change scores indicate improvement in movement dysfunction.
Time Frame: Baseline, Week 8, Week 26, Week 52
Population: Safety Sample - Observed Cases (OC) Data Set and Endpoint - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
units on a scale
  Baseline (n=79, 67, 155, 301) | 0.5 (1.90) | 0.5 (1.02) | 0.3 (1.23) | 0.4 (1.40)
  Change at Week 8 (n=78, 64, 149, 291) | -0.3 (1.45) | -0.1 (0.87) | -0.1 (1.15) | -0.2 (1.18)
  Change at Week 26 (n=61, 49, 130, 240) | -0.4 (1.37) | -0.0 (1.30) | -0.2 (1.26) | -0.2 (1.30)
  Change at Week 52 (n=48, 36, 93, 177) | -0.4 (1.44) | -0.0 (1.00) | -0.1 (1.13) | -0.2 (1.20)
  Change at Endpoint (LOCF) (n=79, 67, 155, 301) | -0.3 (1.33) | 0.0 (1.44) | -0.1 (1.32) | -0.1 (1.35)

4. Primary Outcome: Mean Change From Baseline in Barnes Akathisia Global Clinical Assessment at Week 8, Week 26, Week 52, and Endpoint
Description: The Barnes Akathisia Rating Scale is a 4-item scale to assess presence and severity of drug-induced akathisia, including both objective items and subjective items, together with a global clinical assessment of akathisia. Global assessment is made on a scale of 0 to 5 with comprehensive definitions provided for each anchor point on scale: 0=absent; 1=questionable; 2=mild akathisia; 3=moderate akathisia; 4=marked akathisia; 5=severe akathisia. Score has a possible range from 0 (absent) to 5 (severe akathisia). Negative change scores indicate improvement in akathisia.
Time Frame: Baseline, Week 8, Week 26, Week 52
Population: Safety Sample - Observed Cases (OC) Data Set and Endpoint - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
units on a scale
  Baseline (n=79, 64, 154, 297) | 0.1 (0.57) | 0.2 (0.54) | 0.1 (0.41) | 0.1 (0.49)
  Change at Week 8 (n=78, 60, 149, 287) | -0.1 (0.55) | -0.1 (0.50) | 0.0 (0.35) | 0.0 (0.44)
  Change at Week 26 (n=61, 47, 129, 237) | -0.1 (0.64) | -0.1 (0.48) | 0.0 (0.41) | 0.0 (0.50)
  Change at Week 52 (n=48, 35, 93, 176) | -0.1 (0.37) | 0.0 (0.49) | 0.1 (0.56) | 0.0 (0.50)
  Change at Endpoint (LOCF) (n=79, 64, 154, 297) | 0.0 (0.67) | 0.0 (0.52) | 0.1 (0.58) | 0.0 (0.59)

5. Primary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Metabolic Abnormalities
Description: Abnormal metabolic criterion values include the following: fasting serum glucose ≥115 mg/dL; non-fasting serum glucose ≥ 200 mg/dL; total cholesterol ≥240 mg/dL; LDL cholesterol ≥160 mg/dL; HDL cholesterol ≤30 mg/dL; triglycerides ≥120 mg/dL (females), ≥160 mg/dL (males)
Time Frame: At screening (up to 42 days prior to treatment start), Week 8, Week 26, Week 52
Population: Safety Sample
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Glucose, Fasting Serum | 1 | 1 | 5 | 7
  Glucose, Serum | 0 | 0 | 0 | 0
  Cholesterol, HDL Fasting | 4 | 3 | 7 | 14
  Cholesterol, HDL Non-Fasting | 4 | 3 | 10 | 17
  Cholesterol, HDL Random | 7 | 6 | 16 | 29
  Cholesterol, LDL Fasting | 0 | 0 | 2 | 2
  Cholesterol, LDL Non-Fasting | 0 | 0 | 0 | 0
  Cholesterol, LDL Random | 0 | 0 | 2 | 2
  Cholesterol, Total Fasting | 1 | 0 | 1 | 2
  Cholesterol, Total Non-Fasting | 0 | 0 | 1 | 1
  Cholesterol, Total Random | 1 | 0 | 2 | 3
  Triglycerides, Fasting | 10 | 8 | 20 | 38
  Triglycerides, Non-Fasting | 15 | 12 | 33 | 60
  Triglycerides, Random | 22 | 20 | 47 | 89

6. Primary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Hematology Abnormalities
Description: Abnormal hematology criterion values include the following: hematocrit (ages 6-17, males & females) ≤33%; hemoglobin (ages 6-17, males & females) <11.3 g/dL; leukocytes ≤2800 c/mm3 or ≥16000 c/mm3; eosinophils (ages 6-17, males & females) >17%; neutrophils <15%; platelet count ≤75,000 c/mm3 or ≥700,000 c/mm3
Time Frame: At screening (up to 42 days prior to treatment start), Week 8, Week 26, Week 52
Population: Safety Sample
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Hematocrit | 0 | 0 | 2 | 2
  Hemoglobin | 0 | 2 | 3 | 5
  Leukocytes | 2 | 0 | 3 | 5
  Platelet Count | 0 | 1 | 0 | 1
  Eosinophils, relative | 0 | 1 | 3 | 4
  Neutrophils, relative | 1 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Chemistry Abnormalities
Description: Abnormal chemistry criterion values include the following: aspartate aminotransferase ≥3x upper limit of normal (ULN); alanine aminotransferase ≥3x ULN; alkaline phosphatase ≥3x ULN; lactate dehydrogenase ≥3x ULN; creatinine ≥2.0 mg/dL; uric acid, ≥10.5 mg/dL (male), ≥8.5 mg/dL (female); bilirubin (Total) ≥2.0 mg/dL; serum prolactin >ULN; creatine kinase ≥3x ULN; blood urea nitrogen ≥30 mg/dL; sodium ≤126 mEq/L or ≥156 mEq/L; potassium ≤2.5 mEq/L or ≥ 6.5 mEq/L; chloride ≤90 mEq/L or ≥118 mEq/L; calcium ≤8.2 mg/dL or ≥12 mg/dL
Time Frame: At screening (up to 42 days prior to treatment start), Week 8, Week 26, Week 52
Population: Safety Sample
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Alanine Aminotransferase | 3 | 2 | 5 | 10
  Aspartate Aminotransferase | 0 | 0 | 2 | 2
  Alkaline Phosphatase | 0 | 0 | 0 | 0
  Prolactin | 2 | 0 | 0 | 2
  Lactate Dehydrogenase | 0 | 0 | 0 | 0
  Creatinine | 0 | 0 | 0 | 0
  Uric Acid | 0 | 0 | 0 | 0
  Bilirubin, Total | 0 | 0 | 0 | 0
  Creatine Kinase | 2 | 4 | 7 | 13
  Blood Urea Nitrogen | 0 | 1 | 1 | 2
  Sodium, Serum | 0 | 0 | 0 | 0
  Potassium, Serum | 0 | 0 | 0 | 0
  Chloride, Serum | 0 | 0 | 0 | 0
  Calcium, Total | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Potentially Clinically Relevant Eletrocardiograph (ECG) Abnormalities
Description: These abbreviations are used in the table of ECG measurements: supraventricular (SV), baseline (BL), 1 degree (1°), atrioventricular (A-V), intraventricular (IVT), symmetrical (SYM), corrected QT interval (QTc). QRS complex is a recording of a single heartbeat on ECG corresponding to the depolarization of the right and left ventricles. PR interval is measured from beginning of P wave to beginning of QRS complex. QT interval is a measure of time between start of Q wave and end of T wave in the heart's electrical cycle. ↑ = increase from baseline, ↓ = decrease from baseline, → = "to"
Time Frame: At screening (up to 42 days prior to treatment start), Week 8, Week 26, Week 52
Population: Safety Sample
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Sinus Tachycardia (≥140 bpm & ↑ ≥15 bpm) | 2 | 0 | 2 | 4
  Sinus Bradycardia (≤50 bpm and ↓ ≥15 bpm) | 0 | 0 | 0 | 0
  SV Premature Beat (≥2per10sec & ↑ over BL) | 0 | 0 | 0 | 0
  Ventricular Premature Beat(≥1per10sec & ↑ over BL) | 0 | 0 | 0 | 0
  SV Tachycardia (not present → present) | 0 | 0 | 0 | 0
  Ventricular Tachycardia (not present → present) | 0 | 0 | 0 | 0
  Atrial Fibrillation (not present → present) | 0 | 0 | 0 | 0
  Atrial Flutter (not present → present) | 0 | 0 | 0 | 0
  1° A-V Block (PR ≥ 0.20 sec and ↑ ≥ 0.05 sec) | 0 | 0 | 1 | 1
  2° A-V block (not present → present) | 0 | 0 | 0 | 0
  3° A-V block (not present → present) | 0 | 0 | 0 | 0
  Left Bundle Branch Block (not present → present) | 0 | 0 | 0 | 0
  Right Bundle Branch Block (not present → present) | 0 | 0 | 0 | 0
  Pre-Excitation Syndrome (not present → present) | 0 | 0 | 0 | 0
  Other ITV Block (QRS ≥ 0.10 sec & ↑ 0.02 sec) | 0 | 0 | 3 | 3
  Old Infarction (not present-present at ≥12 weeks) | 0 | 0 | 0 | 0
  Acute/Subacute Infarction (not present → present) | 0 | 0 | 0 | 0
  Myocardial Ischemia (not present → present) | 0 | 0 | 0 | 0
  SYM T-Wave Inversion (not present → present) | 0 | 0 | 0 | 0
  QTcB interval (>475 msec & elevation 10% over BL) | 1 | 0 | 2 | 3
  QTcF interval (>475 msec & elevation 10% over BL) | 1 | 0 | 0 | 1
  Other Abnormality | 3 | 3 | 6 | 12

9. Primary Outcome: Number of Potentially Clinically Relevant Vital Sign Abnormalities
Description: Clinically significantly abnormal vital signs met age-appropriate (heart rate cohorts: ages 5-14 & ages 15+; blood pressure cohorts: ages 6-12 & ages 13-17) criterion AND represented change from pretreatment value of at least the following magnitudes: systolic blood pressure (≥130 mmHg & ≥144 mmHg w/ increase of ≥20 mmHg) or (≤117 mmHg & ≤120 mmHg w/ decrease of ≥20 mmHg); diastolic blood pressure (≥86 mmHg & ≥92 mmHg w/ increase of ≥15 mmHg) or (≤75 mm Hg & ≤80 mmHg w/ decrease of ≥15 mmHg); heart rate (140 bpm and 120 bpm w/ increase of ≥15 bpm) or (50 bpm and 50 bpm w/ decrease of ≥15 bpm).
Time Frame: At screening (up to 42 days prior to treatment start), Week 0 (Baseline), Week 1, Week 2, Week 4, Week 8, Week 14, Week 20, Week 26, Week 34, Week 42, Week 52 (Endpoint)
Population: Safety Sample
Measure: Number; unit: Participants
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Participants
  Supine Systolic Blood Pressure Increase | 5 | 2 | 18 | 25
  Supine Systolic Blood Pressure Decrease | 14 | 15 | 27 | 56
  Standing Systolic Blood Pressure Increase | 6 | 7 | 13 | 26
  Standing Systolic Blood Pressure Decrease | 16 | 22 | 25 | 63
  Sitting Systolic Blood Pressure Increase | 3 | 1 | 6 | 10
  Sitting Systolic Blood Pressure Decrease | 11 | 8 | 13 | 32
  Supine Diastolic Blood Pressure Increase | 6 | 5 | 11 | 22
  Supine Diastolic Blood Pressure Decrease | 15 | 19 | 38 | 72
  Standing Diastolic Blood Pressure Increase | 3 | 8 | 17 | 28
  Standing Diastolic Blood Pressure Decrease | 22 | 20 | 36 | 78
  Sitting Diastolic Blood Pressure Increase | 2 | 2 | 1 | 5
  Sitting Diastolic Blood Pressure Decrease | 14 | 8 | 9 | 31
  Supine Heart Rate Increase | 1 | 1 | 2 | 4
  Supine Heart Rate Decrease | 0 | 0 | 0 | 0
  Standing Heart Rate Increase | 5 | 3 | 4 | 12
  Standing Heart Rate Decrease | 0 | 0 | 1 | 1
  Sitting Heart Rate Increase | 1 | 0 | 1 | 2
  Sitting Heart Rate Decrease | 0 | 0 | 0 | 0

10. Primary Outcome: Mean Change From Baseline in Patient Weight
Time Frame: as for outcome 9
Population: Safety Sample - Observed Cases (OC) Data Set and Endpoint - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
kg
  Baseline (n=84, 69, 169, 322) | 42.5 (23.17) | 45.1 (20.37) | 45.4 (21.79) | 44.6 (21.83)
  Change at Week 1 (n=78, 58, 149, 285) | 0.2 (0.76) | -0.1 (1.06) | 0.4 (0.94) | 0.3 (0.94)
  Change at Week 2 (n=81, 67, 165, 313) | 0.2 (0.99) | 0.0 (1.47) | 0.8 (1.15) | 0.5 (1.23)
  Change at Week 4 (n=80, 67, 165, 312) | 0.8 (1.26) | 0.5 (1.60) | 1.2 (1.43) | 1.0 (1.45)
  Change at Week 8 (n=77, 65, 149, 291) | 1.6 (1.99) | 1.5 (2.29) | 1.9 (2.09) | 1.8 (2.11)
  Change at Week 14 (n=71, 55, 142, 268) | 3.3 (2.81) | 2.8 (2.79) | 3.1 (2.80) | 3.1 (2.80)
  Change at Week 20 (n=66, 50, 136, 252) | 4.0 (3.39) | 3.3 (4.73) | 4.2 (3.34) | 4.0 (3.67)
  Change at Week 26 (n=61, 49, 130, 240) | 5.0 (4.41) | 4.7 (4.36) | 4.9 (3.99) | 4.9 (4.16)
  Change at Week 34 (n=60, 46, 123, 229) | 6.0 (5.80) | 5.8 (4.90) | 6.1 (4.68) | 6.0 (5.02)
  Change at Week 42 (n=58, 43, 115, 216) | 7.0 (6.46) | 6.4 (5.90) | 7.1 (5.11) | 6.9 (5.64)
  Change at Week 52 (n=48, 36, 94, 178) | 8.7 (6.77) | 7.7 (6.44) | 7.9 (5.90) | 8.1 (6.23)
  Change at Endpoint (LOCF) (n=84, 69, 169, 322) | 6.3 (6.71) | 5.5 (5.50) | 6.6 (5.72) | 6.3 (5.94)

11. Primary Outcome: Mean Change From Baseline by Time Period in Body Weight Z-Score
Description: The Z-Score indicates how many standard deviations a person is from the population norm values. The body weight z-scores are designed to take into account the amount of weight gain that would be expected due to normal growth in children and adolescents. The body weight z-scores are by age and gender standardized values (corresponding to a normal distribution with mean 0 and a standard deviation of 1) of the actual weight measurements, based on the Growth Charts provided by the Centers for Disease Control (CDC; see Links section of this record).
Time Frame: as for outcome 9
Population: Safety Sample. Subjects included in the period evaluation had a baseline and at least 1 measurement within the time period that was assessed. Patients are only counted once in each time period but can appear in multiple time periods. For those with multiple records in 1 time period, only the last record in that period is included in calculations.
Measure: Mean (Standard Deviation); unit: Standard Deviations away from Population
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Standard Deviations away from Population
  Baseline (n=84, 70, 169, 323) | 0.47 (1.687) | 0.95 (1.112) | 0.98 (1.392) | 0.84 (1.434)
  <= 3 Months (n=84, 70, 169, 323) | 0.13 (0.283) | 0.10 (0.204) | 0.09 (0.300) | 0.10 (0.277)
  3-6 Months (n=73, 56, 145, 274) | 0.24 (0.433) | 0.26 (0.331) | 0.20 (0.327) | 0.22 (0.359)
  6-9 Months (n=63, 49, 131, 243) | 0.31 (0.570) | 0.28 (0.367) | 0.23 (0.407) | 0.26 (0.448)
  >9 Months (n=59, 44, 115, 218) | 0.33 (0.580) | 0.23 (0.399) | 0.24 (0.465) | 0.26 (0.486)

12. Primary Outcome: Mean Change From Baseline in Patient Body Mass Index (BMI)
Description: The body mass index (BMI) is a statistical measurement which compares a person's weight and height. Though it does not actually measure the percentage of body fat, it is used to estimate a healthy body weight based on subject height.
Time Frame: as for outcome 9
Population: Safety Sample: Endpoint - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
kg/m2
  Baseline (n=84, 69, 169, 322) | 20.1 (6.31) | 21.0 (5.15) | 21.6 (6.38) | 21.1 (6.13)
  Change at Endpoint (LOCF) (n=84, 69, 169, 322) | 1.7 (2.56) | 1.4 (2.07) | 1.8 (2.51) | 1.7 (2.43)

13. Primary Outcome: Mean Change From Baseline By Time Period in BMI Z-Score
Description: The Z-Score indicates how many standard deviations a person is from the population norm values. The BMI z-scores are designed to take into account the BMI that would be expected due to normal growth in children and adolescents. The BMI z-scores are by age and gender standardized values (corresponding to a normal distribution with mean 0 and a standard deviation of 1) of the actual BMI measurements, based on the Growth Charts provided by the Centers for Disease Control (CDC; see Links section of this record).
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Standard Deviations away from Population
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
Standard Deviations away from Population
  Baseline (n=84, 70, 169, 323) | 0.44 (1.591) | 0.98 (0.997) | 1.01 (1.236) | 0.86 (1.313)
  <=3 Months (n=84, 70, 169, 323) | 0.17 (0.436) | 0.12 (0.268) | 0.09 (0.500) | 0.12 (0.443)
  3-6 Months (n=73, 56, 145, 274) | 0.29 (0.625) | 0.28 (0.388) | 0.18 (0.549) | 0.23 (0.543)
  6-9 Months (n=62, 49, 129, 240) | 0.36 (0.647) | 0.24 (0.438) | 0.18 (0.643) | 0.24 (0.611)
  >9 Months (n=59, 44, 115, 218) | 0.33 (0.768) | 0.15 (0.476) | 0.14 (0.775) | 0.19 (0.725)

14. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression (CGI)-Severity Score at Week 52 (Endpoint, LOCF)
Description: CGI scale is a global evaluation of improvement over time. CGI-Severity (CGI-S) is a clinician-rated assessment that evaluates the severity of a patient's condition on a 7-point scale ranging from 1 (no symptoms) to 7 (very severe symptoms). CGI-Severity score is from 1 to 7. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: Efficacy Sample, LOCF. The Efficacy Sample includes all patients that had a baseline and at least one post-baseline measurement of the same scale. A total of 322 patients met this criterion based on CGI-S evaluations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 84 | 69 | 169 | 322
units on a scale
  Baseline | 4.8 (0.99) | 4.2 (0.99) | 3.9 (1.05) | 4.2 (1.08)
  Change at Endpoint (LOCF) | -0.8 (0.85) | -0.4 (1.06) | -0.0 (1.01) | -0.3 (1.04)

15. Secondary Outcome: CGI-Improvement Score at Week 52 (Endpoint, LOCF)
Description: CGI scale is a global evaluation of improvement over time. CGI-Improvement (CGI-I) is a clinician rated assessment that evaluates improvement relative to symptoms at baseline on a a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). CGI-I Score is from 1 to 7. A lower score signifies larger improvement.
Time Frame: Week 52 (Endpoint, LOCF)
Population: Efficacy Sample. The Efficacy Sample includes all patients that had a baseline and at least one post-baseline measurement of the same scale. A total of 322 patients met this criterion based on CGI-S evaluations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 84 | 69 | 169 | 322
units on a scale | 2.7 (1.30) | 2.4 (1.24) | 2.5 (1.20) | 2.5 (1.23)

16. Secondary Outcome: Mean Change From Baseline in Aberrant Behavior Checklist (ABC) Irritability Score at Week 52 (Endpoint, LOCF)
Description: The ABC is an informant-based symptom checklist for assessing and classifying problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0 = not at all a problem to 3 = the problem is severe in degree), and resolve into 5 subscales: (1) irritability and agitation; (2) lethargy and social withdrawal; (3) stereotypic behavior; (4) hyperactivity and noncompliance, and (5) inappropriate speech. ABC Irritability Subscale Score is from 0 to 45. A negative change signifies improvement
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: Efficacy Sample, LOCF. The Efficacy Sample includes all patients that had a baseline and at least one post-baseline measurement of the same scale. A total of 322 patients met this criterion based on CGI-S evaluations. Of those, 8 patients had baseline ABC (all subscales) evaluations but no post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 80 | 68 | 166 | 314
units on a scale
  Baseline | 23.2 (8.88) | 21.5 (9.82) | 15.0 (9.20) | 18.5 (9.96)
  Change at Endpoint (LOCF) | -6.5 (11.12) | -6.1 (11.25) | 0.7 (9.72) | -2.6 (10.98)

17. Secondary Outcome: Mean Change From Baseline in ABC Hyperactivity Subscale Score at Week 52 (Endpoint, LOCF)
Description: The ABC is an informant-based symptom checklist for assessing and classifying problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0 = not at all a problem to 3 = the problem is severe in degree), and resolve into 5 subscales: (1) irritability and agitation; (2) lethargy and social withdrawal; (3) stereotypic behavior; (4) hyperactivity and noncompliance, and (5) inappropriate speech. ABC Hyperactivity Subscale Score is from 0 to 48. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: Efficacy Sample, LOCF.The Efficacy Sample includes all patients that had a baseline and at least one post-baseline measurement of the same scale. A total of 322 patients met this criterion based on CGI-S evaluations. Of those, 8 patients had baseline ABC (all subscales) evaluations but no post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 80 | 68 | 166 | 314
units on a scale
  Baseline | 28.4 (10.87) | 25.8 (13.18) | 18.4 (12.03) | 22.5 (12.79)
  Change at Endpoint (LOCF) | -10.0 (10.55) | -8.3 (10.85) | 0.3 (11.18) | -4.2 (11.92)

18. Secondary Outcome: Change From Baseline in ABC Stereotypy Subscale Score at Week 52 (Endpoint, LOCF)
Description: The ABC is an informant-based symptom checklist for assessing and classifying problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0 = not at all a problem to 3 = the problem is severe in degree), and resolve into 5 subscales: (1) irritability and agitation; (2) lethargy and social withdrawal; (3) stereotypic behavior; (4) hyperactivity and noncompliance, and (5) inappropriate speech. ABC Stereotypy Subscale Score is from 0 to 21. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 80 | 68 | 166 | 314
units on a scale
  Baseline | 8.1 (5.18) | 8.1 (5.57) | 6.4 (5.46) | 7.2 (5.46)
  Change at Endpoint (LOCF) | -2.5 (4.67) | -1.9 (4.46) | 0.1 (4.58) | -1.0 (4.71)

19. Secondary Outcome: Mean Change From Baseline in ABC Social Withdrawal Scale At Week 52 (Endpoint, LOCF)
Description: The ABC is an informant-based symptom checklist for assessing and classifying problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0 = not at all a problem to 3 = the problem is severe in degree), and resolve into 5 subscales: (1) irritability and agitation; (2) lethargy and social withdrawal; (3) stereotypic behavior; (4) hyperactivity and noncompliance, and (5) inappropriate speech. ABC Social Withdrawal Subscale Score is from 0 to 48. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 80 | 68 | 166 | 314
units on a scale
  Baseline | 14.6 (8.62) | 11.3 (9.24) | 10.4 (8.86) | 11.7 (9.03)
  Change at Endpoint (LOCF) | -5.4 (9.07) | -3.0 (6.96) | -1.8 (6.09) | -3.0 (7.28)

20. Secondary Outcome: Mean Change From Baseline in ABC Inappropriate Speech Subscale Score at Week 52 (Endpoint, LOCF)
Description: The ABC is an informant-based symptom checklist for assessing and classifying problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0 = not at all a problem to 3 = the problem is severe in degree), and resolve into 5 subscales: (1) irritability and agitation; (2) lethargy and social withdrawal; (3) stereotypic behavior; (4) hyperactivity and noncompliance, and (5) inappropriate speech. ABC Inappropriate Speech Subscale score is from 1 to 12. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: Efficacy Sample, LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 86 | 70 | 174 | 330
units on a scale
  Baseline | 5.8 (3.15) | 5.7 (4.23) | 4.2 (3.61) | 4.9 (3.72)
  Change at Endpoint (LOCF) | -1.9 (2.66) | -1.8 (2.94) | -0.3 (2.50) | -1.0 (2.75)

21. Secondary Outcome: Change From Baseline in Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) Score at Week 52 (Endpoint, LOCF)
Description: CY-BOCS is a 10-item, clinician-rated scale designed to measure the severity of obsessive-compulsive symptoms in patients below the age of 18. The scale contains 5 items pertaining to obsessions (which were not used in this trial) and 5 items pertaining to compulsions, which rated each symptom domain in terms of time spent, interference with functioning, distress, resistance, and control. Each item was rated on a 5-point scale, from 0 (no symptoms or minimum severity) to 4 (extreme symptoms or maximum severity). CY-BOCS Score is from 0 to 20. A negative change score signifies improvement.
Time Frame: Week 0 (Baseline), Week 52 (Endpoint, LOCF)
Population: Efficacy Sample, LOCF. The Efficacy Sample includes all patients that had a baseline and at least one post-baseline measurement of the same scale. A total of 322 patients met this criterion based on CGI-S evaluations. Of those, 96 patients did not have post-baseline evaluations for CY-BOCS, and were excluded from the efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo | Rollover Placebo | Rollover Aripiprazole | Total
Number analyzed (Participants) | 62 | 49 | 115 | 226
units on a scale
  Baseline | 12.6 (4.60) | 12.1 (3.96) | 10.4 (3.87) | 11.4 (4.20)
  Change at Endpoint (LOCF) | -2.0 (3.68) | -2.4 (5.06) | 0.2 (3.81) | -0.9 (4.23)

ADVERSE EVENTS:
Arm/Group | De Novo | Roll Over Aripiprazole | Roll Over Placebo
Serious Adverse Events (participants affected / at risk) | 3/86 | 5/174 | 1/70
Other Adverse Events (participants affected / at risk) | 73/86 | 136/174 | 61/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=86) | Roll Over Aripiprazole (N=174) | Roll Over Placebo (N=70)
AGGRESSION (Psychiatric disorders) | 1 | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0 | 0
IMPULSIVE BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 0 | 1 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=86) | Roll Over Aripiprazole (N=174) | Roll Over Placebo (N=70)
WEIGHT INCREASED (Investigations) | 20 | 40 | 16
TIC (Psychiatric disorders) | 0 | 2 | 6
ANXIETY (Psychiatric disorders) | 3 | 10 | 0
INSOMNIA (Psychiatric disorders) | 8 | 17 | 8
AGITATION (Psychiatric disorders) | 8 | 11 | 2
AGGRESSION (Psychiatric disorders) | 8 | 15 | 6
DROOLING (Nervous system disorders) | 3 | 16 | 3
HEADACHE (Nervous system disorders) | 7 | 18 | 7
LETHARGY (Nervous system disorders) | 7 | 2 | 1
SEDATION (Nervous system disorders) | 8 | 9 | 10
DYSKINESIA (Nervous system disorders) | 5 | 3 | 0
SOMNOLENCE (Nervous system disorders) | 4 | 3 | 6
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 4
VOMITING (Gastrointestinal disorders) | 17 | 34 | 11
DIARRHOEA (Gastrointestinal disorders) | 7 | 15 | 8
CONSTIPATION (Gastrointestinal disorders) | 6 | 7 | 4
SINUSITIS (Infections and infestations) | 7 | 10 | 2
EAR INFECTION (Infections and infestations) | 3 | 15 | 2
NASOPHARYNGITIS (Infections and infestations) | 12 | 22 | 10
GASTROENTERITIS VIRAL (Infections and infestations) | 5 | 8 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 16 | 11
ENURESIS (Renal and urinary disorders) | 5 | 6 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 7 | 2
INCREASED APPETITE (Metabolism and nutrition disorders) | 16 | 19 | 8
RASH (Skin and subcutaneous tissue disorders) | 5 | 7 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 6
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
FATIGUE (General disorders) | 7 | 9 | 7
PYREXIA (General disorders) | 6 | 23 | 10
IRRITABILITY (General disorders) | 4 | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.